CLINICAL TRIAL: NCT03299101
Title: Pilot Testing a Home-based Rehabilitation Intervention Designed to Improve Outcomes of Frail Veterans Following Cardiothoracic Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: E2562-P; I21RX002562 (NIH)
Record Dates: First submitted 2017-09-18; First posted 2017-10-02 (Actual); Results first posted 2020-12-21 (Actual); Last update posted 2021-01-13 (Actual); Status verified 2020-12

CONDITIONS: Coronary Artery Bypass Graft; Non-cardiac Thoracic Surgery; Frailty
Keywords: Frailty; Prehabilitation; Exercise therapy; Surgery; Nutrition support
MeSH Terms: conditions — Frailty | interventions — Preoperative Exercise

STUDY DESIGN:
Intervention Model Description: A novel a novel, multifaceted, home-based prehabilitation intervention designed to improve functional capacity and postoperative outcomes for frail Veterans anticipating cardiothoracic surgery. Prehabilitation will include: (a) aerobic conditioning; (b) strength and coordination training; (c) respiratory muscle training; and (d) nutritional coaching and supplementation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Prehabilitation (Experimental): Prospective sample of patients anticipating cardiothoracic surgery.
  Interventions: Other: Prehabilitation

INTERVENTIONS:
Other: Prehabilitation — Prehabilitation will last 4 weeks and consist of a novel, home-based regimen of (a) aerobic conditioning; (b) strength and coordination training; (c) respiratory muscle training; and (d) nutritional coaching and supplementation.

SUMMARY:
Frail Veterans are at increased risk for poor surgical outcomes, and as the Veteran population grows older and more frail, there is a critical need to identify effective strategies for reducing surgical risks for these patients. Prior research shows that inter-disciplinary rehabilitation strategies deployed after surgery enhance recovery and improve outcomes by building strength and improving nutrition. The investigators believe that similar improvements may be obtained by using similar interventions before surgery to "prehabilitate" patients' capacity to tolerate the stress of surgery. The proposed research will examine the feasibility of a new, home-based prehabilitation intervention aimed at improving surgical outcomes after cardiothoracic surgery through preoperative exercise training and nutritional supplementation. Findings from the study will inform the design of a larger randomized controlled trial of the prehabilitation intervention. If proven effective, prehabilitation could benefit as many as 42,000 frail Veterans who are scheduled for major elective surgery each year.

DETAILED DESCRIPTION:
Background: Frail Veterans are at increased risk for poor surgical outcomes. Although surgical techniques have advanced to a level where surgery on very old adults is feasible, if a patient is also frail, the stress of surgery may overwhelm their adaptive capacities, placing them at increased risk of mortality, morbidity, and institutionalization even if surgery is technically successful. Frailty is a clinical syndrome that is commonly characterized by muscle atrophy, diminished strength and speed, decreased physical activity, and exhaustion. It is independent of any specific disease, but it increases with age and worsens disease prognoses by diminishing capacity to tolerate stressors. Thus, while surgery is often indicated for older patients, frail candidates are less likely than robust counterparts to tolerate the procedure and/or recover functional capacity. In fact, recent VA data demonstrate that frailty is a more powerful predictor of increased perioperative mortality, morbidity, length of stay, and cost than predictions based on age or comorbidity alone. As the Veteran and US populations grow older, frailty will increase, making it critically important to identify effective strategies for improving the surgical recovery and outcomes of frail patients.

"Prehabilitation" has the potential to improve surgical outcomes among the frail. Prior research demonstrates that inter-disciplinary rehabilitation strategies deployed after surgery enhance recovery and improve outcomes by building strength and improving nutrition. Based on this success, there is growing interest in "prehabilitation", which is a similar intervention deployed before surgery. By modifying physiological and environmental risks, prehabilitation aims to augment patients' capacity to compensate for the stress of surgery itself and the convalescent period thereafter. Frail patients may benefit disproportionately from prehabilitation because they have diminished capacity to endure the procedure and/or recovery. Preliminary evidence suggests that preoperative exercise interventions improve surgical outcomes. However, prehabilitation has not yet been studied in either Veteran or specifically frail populations, and no prior studies used home-based prehabilitation strategies to safely minimize travel-related barriers to participation.

Objectives: The investigators will examine the feasibility of a novel, multifaceted, home-based prehabilitation intervention designed to improve functional capacity and postoperative outcomes for frail Veterans anticipating cardiothoracic surgery. Specific aims are to:

1. Estimate rates of recruitment, retention, and adherence to the intervention; and evaluate participation barriers.
2. Measure changes over time in frailty, physical function, pulmonary function, nutrition, and health-related quality of life at baseline, the day of surgery, and 30 and 90 days after surgery.
3. Explore changes in postoperative mortality, major complications, length of hospital stay, and level of independent living using case-matched historical controls.

Methods: This single-arm pilot study will enroll a consecutive cohort of up to 50 Veterans identified as frail using a standardized frailty assessment and scheduled for major cardiothoracic surgery at the VA Pittsburgh Healthcare System. The 4 week long prehabilitation regimen will include: (a) aerobic conditioning, (b) strength and coordination training, (c) respiratory muscle training, and (d) nutritional coaching and supplementation. Pre- and post-prehabilitation assessments will include: (a) frailty; (b) physical function; (c) pulmonary function; (d) nutrition; and (e) health-related quality of life. Postoperative outcomes will include length of stay, mortality and complications. Compliance with the prehabilitation regimen will be assessed through patient logs and pedometers. Analyses will inform a larger randomized controlled trial testing the prehabilitation intervention. Findings will be relevant for the 42,000 frail Veterans scheduled for major elective surgery each year.

ELIGIBILITY:
Inclusion Criteria:

1. Veteran patient scheduled for Coronary artery bypass graft (CABG), valve surgery, or other non-cardiac thoracic surgery;
2. Demonstrate at least mild frailty (e.g., Risk Analysis Index [RAI]>=16).
3. Physician/provider request for patients with RAI<16.

Exclusion Criteria:

* Emergent, urgent, or otherwise time-sensitive surgery that precludes prehabilitation;
* Unstable or recent unstable cardiac syndrome as defined by (a) acute coronary syndrome within 6 weeks; (b) decompensated heart failure; (c) New York Heart Association Class IV Heart Failure; (d) unstable angina; (e) Canadian Cardiovascular Society Class IV symptoms; (f) critical left main coronary disease; (g) clinically significant arrhythmias,
* Severe valvular heart disease: (a) severe aortic or mitral stenosis (aortic or mitral valve area <1.0 cm2 or mean gradient >40 or >10 mm Hg, respectively)
* Dynamic LV (Left Ventricle) outflow obstruction
* Physical, cognitive, social or logistical limitations preventing participation in the prehabilitation regimen, including:
* Patients who require surrogate consent for the planned surgery
* Patients with court orders of incompetence or clinical determinations of incapacity documented in the medical record
* Clinical exam by study physician consistent with incapacity
* Patients who at any time during prehabilitation or longitudinal follow up demonstrate insufficient cognitive capacity to safely and effectively carry out the prescribed activities.
* Unable to speak English.
* Surgery is cancelled by IMPACT clinic or surgeon due to unacceptable risk.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2017-11-22 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2020-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel E. Hall, MD MDiv MHSc, Principal Investigator — VA Pittsburgh Healthcare System University Drive Division, Pittsburgh, PA
Locations (1):
- VA Pittsburgh Healthcare System University Drive Division, Pittsburgh, PA, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Prehabilitation
Started | 35
Completed | 25
Not Completed | 10
Not completed — Lost to Follow-up | 1
Not completed — Withdrawal by Subject | 5
Not completed — Surgery was changed | 3
Not completed — Not enough time to complete prehab | 1

BASELINE CHARACTERISTICS:
Population: All participants that completed the baseline assessments were analyzed.
Arm/Group | Prehabilitation
Number analyzed (Participants) | 33
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 11
  >=65 years | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.09 (7.66)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 31
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 33
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 31
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 33
Risk Analysis Index [Mean (Standard Deviation); unit: Score on a scale] — This recently published frailty index is assessed by a clinician administered questionnaire. The score and reflects frailty-associated mortality risk ranging from 0-81. Higher scores indicate higher risk for post operative complications and other frailty-related outcomes.
  Score on a scale | 17.85 (8.92)

OUTCOME MEASURES:

1. Primary Outcome: Recruitment Rate
Description: Recruitment will be expressed as the percentage of eligible patients approached who agree to participate in this pilot study.
Time Frame: Baseline
Population: 65 is the number of patients approached.
Measure: Count of Participants; unit: Participants
Arm/Group | Prehabilitation
Number analyzed (Participants) | 65
Participants | 35

2. Primary Outcome: Retention Rate
Description: Retention rate will be expressed as the percentage of enrolled patients who were retained in the study and completed study procedures. It will be calculated for incremental steps along the study timeline and at the completion of study procedures 90 days postoperatively.
Time Frame: 90 days postoperatively
Measure: Count of Participants; unit: Participants
Arm/Group | Prehabilitation
Number analyzed (Participants) | 35
Participants | 25

3. Primary Outcome: Adherence Rate
Description: Compliance rates will be expressed as the percentage of assigned activities actually completed by patients as recorded in home exercise and nutrition logs.
Time Frame: Day of surgery
Population: All participants that self-reported their home training and/or showed their exercise or nutrition logs were analyzed.
Measure: Mean (Standard Deviation); unit: percentage of activities completed
Arm/Group | Prehabilitation
Number analyzed (Participants) | 27
percentage of activities completed
  Home Strength/Aerobic/Transition Training: number analyzed (Participants) | 26
  Home Strength/Aerobic/Transition Training | 78.85 (28.96)
  Home Breathing Training | 86.30 (24.20)
  Home Nutrition Log: number analyzed (Participants) | 22
  Home Nutrition Log | 64.09 (14.10)

4. Secondary Outcome: Change in Grip Strength Over the Course of Treatment and Recovery.
Description: Grip strength will be measured in kilograms of pressure using a Smedley grip dynamometer
Time Frame: Baseline, day of surgery, 90 days postoperatively
Population: All participants that completed the hand grip assessment were analyzed at each completed timepoint.
Measure: Mean (Standard Deviation); unit: kgf/cm2
Arm/Group | Prehabilitation
Number analyzed (Participants) | 33
kgf/cm2
  Baseline Grip Strength | 31.52 (9.27)
  Day of Surgery Grip Strength: number analyzed (Participants) | 25
  Day of Surgery Grip Strength | 32.19 (7.89)
  90 Days Post Surgery: number analyzed (Participants) | 22
  90 Days Post Surgery | 31.13 (9.99)
Statistical Analysis 1: Comparison: Prehabilitation; Linear mixed models estimated overall, within-person change in grip strength across all 4 time points; Test type: Superiority; p = 0.872, Mixed Models Analysis
Statistical Analysis 2: Comparison: Prehabilitation; Linear mixed models estimated within-person change in grip strength between baseline and day of surgery; Test type: Superiority; p = 0.423, Mixed Models Analysis — The null hypothesis was rejected a priori if p<.05; Mean Difference (Net) = 0.57, Standard Error of Mean 0.71 — The mean within-person difference was assessed with linear mixed models with standard error and p-value similar to paired t-tests
Statistical Analysis 3: Comparison: Prehabilitation; Linear mixed models estimated within-person change in grip strength between baseline and 90 days postop; Test type: Superiority; p = 0.853, Mixed Models Analysis — The null hypothesis was rejected a priori if p<.05; Mean Difference (Net) = -0.39, Standard Error of Mean 2.12 — [estimate comment as in outcome 4, analysis 2]
Statistical Analysis 4: Comparison: Prehabilitation; Linear mixed models estimated within-person change in grip strength between day of surgery and 90 days postop; Test type: Superiority; p = 0.552, Mixed Models Analysis — The null hypothesis was rejected a priori if p<.05; Mean Difference (Net) = -1.28, Standard Error of Mean 2.16 — [estimate comment as in outcome 4, analysis 2]

5. Secondary Outcome: Change in Pulmonary Function Over the Course of Treatment and Recovery: Max MIP
Description: Pulmonary function will be measured in terms of maximum MIP (maximal inspiratory pressure).
Time Frame: Baseline, day of surgery, 90 days postoperatively
Population: All participants that completed the pulmonary function assessments were analyzed at each completed timepoint.
Measure: Mean (Standard Deviation); unit: cm of H2O
Arm/Group | Prehabilitation
Number analyzed (Participants) | 33
cm of H2O
  Baseline Max MIP | 71.42 (24.54)
  Day of surgery Max MIP: number analyzed (Participants) | 26
  Day of surgery Max MIP | 77.96 (24.23)
  90 Day Postop Max MIP: number analyzed (Participants) | 22
  90 Day Postop Max MIP | 79.82 (26.86)
Statistical Analysis 1: Comparison: Prehabilitation; Linear mixed models estimated overall, within-person change in max MIP across all 4 time points; Test type: Superiority; p = 0.256, Mixed Models Analysis — The null hypothesis was rejected a priori if p<.05
Statistical Analysis 2: Comparison: Prehabilitation; Linear mixed models estimated within-person change in maximum MIP between baseline and day of surgery; Test type: Superiority; p = 0.091, Mixed Models Analysis — The null hypothesis was rejected a priori if p<.05; Mean Difference (Net) = 4.69, Standard Error of Mean 2.78 — [estimate comment as in outcome 4, analysis 2]
Statistical Analysis 3: Comparison: Prehabilitation; Linear mixed models estimated within-person change in maximum MIP between baseline and 90 days postop; Test type: Superiority; p = 0.066, Mixed Models Analysis — The null hypothesis was rejected a priori if p<.05; Mean Difference (Net) = 6.80, Standard Error of Mean 3.69 — [estimate comment as in outcome 4, analysis 2]
Statistical Analysis 4: Comparison: Prehabilitation; Linear mixed models estimated within-person change in maximum MIP between day of surgery and 90 days postop; Test type: Superiority; p = 0.552, Mixed Models Analysis — The null hypothesis was rejected a priori if p<.05; Mean Difference (Net) = 1.86, Standard Error of Mean 3.13 — [estimate comment as in outcome 4, analysis 2]

6. Secondary Outcome: Change in Pulmonary Function Over the Course of Treatment and Recovery: Mean MIP
Description: Pulmonary function will be measured in terms of mean maximal inspiratory pressure (MIP).
Time Frame: Baseline, day of surgery, 90 days postoperatively
Population: All participants that completed the pulmonary function assessments were analyzed at each completed timepoint.
Measure: Mean (Standard Deviation); unit: cm of H2O
Arm/Group | Prehabilitation
Number analyzed (Participants) | 33
cm of H2O
  Baseline Mean MIP | 60.69 (23.57)
  Day of surgery Mean MIP: number analyzed (Participants) | 26
  Day of surgery Mean MIP | 69.38 (23.11)
  90 Day Postop Mean MIP: number analyzed (Participants) | 22
  90 Day Postop Mean MIP | 71.43 (26.10)
Statistical Analysis 1: Comparison: Prehabilitation; Linear mixed models estimated overall, within-person change in mean MIP across all 4 time points; Test type: Superiority; p = 0.003, Mixed Models Analysis — The null hypothesis was rejected a priori if p<.05
Statistical Analysis 2: Comparison: Prehabilitation; Linear mixed models estimated within-person change in mean MIP between baseline and day of surgery; Test type: Superiority; p = 0.003, Mixed Models Analysis — The null hypothesis was rejected a priori if p<.05; Mean Difference (Net) = 7.48, Standard Error of Mean 2.48 — [estimate comment as in outcome 4, analysis 2]
Statistical Analysis 3: Comparison: Prehabilitation; Linear mixed models estimated within-person change in mean MIP between baseline and 90 days postop; Test type: Superiority; p = 0.005, Mixed Models Analysis — The null hypothesis was rejected a priori if p<.05; Mean Difference (Net) = 10.18, Standard Error of Mean 3.61 — [estimate comment as in outcome 4, analysis 2]
Statistical Analysis 4: Comparison: Prehabilitation; Linear mixed models estimated within-person change in mean MIP between day of surgery and 90 days postop; Test type: Superiority; p = 0.290, Mixed Models Analysis — The null hypothesis was rejected a priori if p<.05; Mean Difference (Net) = 2.31, Standard Error of Mean 2.18 — [estimate comment as in outcome 4, analysis 2]

7. Secondary Outcome: Change in Pulmonary Function Over the Course of Treatment and Recovery: Max MEP
Description: Pulmonary function will be measured in terms of maximum MEP (maximal expiratory pressures)
Time Frame: Baseline, day of surgery, 90 days postoperatively
Population: All participants that completed the pulmonary function assessments were analyzed at each completed timepoint.
Measure: Mean (Standard Deviation); unit: cm of H2O
Arm/Group | Prehabilitation
Number analyzed (Participants) | 33
cm of H2O
  Baseline Max MEP | 108.09 (33.64)
  Day of surgery Max MEP: number analyzed (Participants) | 26
  Day of surgery Max MEP | 120.81 (30.40)
  90 Day Postop Max MEP: number analyzed (Participants) | 22
  90 Day Postop Max MEP | 123.64 (32.64)
Statistical Analysis 1: Comparison: Prehabilitation; Linear mixed models estimated overall, within-person change in maximal inspiratory pressure across all 4 time points; Test type: Superiority; p = 0.009, Mixed Models Analysis — The null hypothesis was rejected a priori if p<.05
Statistical Analysis 2: Comparison: Prehabilitation; Linear mixed models estimated within-person change in maximum MEP between baseline and day of surgery; Test type: Superiority; p = 0.006, Mixed Models Analysis — The null hypothesis was rejected a priori if p<.05; Mean Difference (Net) = 12.61, Standard Error of Mean 4.57 — [estimate comment as in outcome 4, analysis 2]
Statistical Analysis 3: Comparison: Prehabilitation; Linear mixed models estimated within-person change in maximum MEP between baseline and 90 days postop; Test type: Superiority; p = 0.015, Mixed Models Analysis — The null hypothesis was rejected a priori if p<.05; Mean Difference (Net) = 12.79, Standard Error of Mean 5.25 — [estimate comment as in outcome 4, analysis 2]
Statistical Analysis 4: Comparison: Prehabilitation; Linear mixed models estimated within-person change in maximum MEP between day of surgery and 90 days postop; Test type: Superiority; p = 0.802, Mixed Models Analysis — The null hypothesis was rejected a priori if p<.05; Mean Difference (Net) = -0.86, Standard Error of Mean 3.42 — [estimate comment as in outcome 4, analysis 2]

8. Secondary Outcome: Change in Pulmonary Function Over the Course of Treatment and Recovery: Mean MEP
Description: Pulmonary function will be measured in terms of mean maximal expiratory pressures (MEP).
Time Frame: Baseline, day of surgery, 90 days postoperatively
Population: All participants that completed the pulmonary function assessments were analyzed at each completed timepoint.
Measure: Mean (Standard Deviation); unit: cm of H2O
Arm/Group | Prehabilitation
Number analyzed (Participants) | 33
cm of H2O
  Baseline Mean MEP | 98.48 (32.90)
  Day of surgery Mean MEP: number analyzed (Participants) | 26
  Day of surgery Mean MEP | 111.22 (28.62)
  90 Day Postop Mean MEP: number analyzed (Participants) | 22
  90 Day Postop Mean MEP | 112.01 (31.72)
Statistical Analysis 1: Comparison: Prehabilitation; Linear mixed models estimated overall, within-person change in Mean MEP across all 4 time points; Test type: Superiority; p = 0.010, Mixed Models Analysis — The null hypothesis was rejected a priori if p<.05
Statistical Analysis 2: Comparison: Prehabilitation; Linear mixed models estimated within-person change in mean MEP between baseline and day of surgery; Test type: Superiority; p = 0.004, Mixed Models Analysis — The null hypothesis was rejected a priori if p<.05; Mean Difference (Net) = 12.37, Standard Error of Mean 4.35 — [estimate comment as in outcome 4, analysis 2]
Statistical Analysis 3: Comparison: Prehabilitation; Linear mixed models estimated within-person change in mean MEP between baseline and 90 days postop; Test type: Superiority; p = 0.042, Mixed Models Analysis — The null hypothesis was rejected a priori if p<.05; Mean Difference (Net) = 9.95, Standard Error of Mean 4.90 — [estimate comment as in outcome 4, analysis 2]
Statistical Analysis 4: Comparison: Prehabilitation; Linear mixed models estimated within-person change in mean MEP between day of surgery and 90 days postop; Test type: Superiority; p = 0.221, Mixed Models Analysis — The null hypothesis was rejected a priori if p<.05; Mean Difference (Net) = -3.77, Standard Error of Mean 3.08 — [estimate comment as in outcome 4, analysis 2]

9. Secondary Outcome: Change in Pulmonary Function Over the Course of Treatment and Recovery: Max SMIP
Description: Pulmonary function will be measured in terms of maximum sustained MIP (SMIP).
Time Frame: Baseline, day of surgery, 90 days postoperatively
Population: All participants that completed the pulmonary function assessments were analyzed at each completed timepoint.
Measure: Mean (Standard Deviation); unit: cm of H2O
Arm/Group | Prehabilitation
Number analyzed (Participants) | 33
cm of H2O
  Baseline Max SMIP | 416.55 (197.85)
  Day of surgery Max SMIP: number analyzed (Participants) | 25
  Day of surgery Max SMIP | 434.48 (192.42)
  90 Day Postop Max SMIP: number analyzed (Participants) | 22
  90 Day Postop Max SMIP | 466.77 (197.27)
Statistical Analysis 1: Comparison: Prehabilitation; Linear mixed models estimated overall, within-person change in max SMIP across all 4 time points; Test type: Superiority; p = 0.814, Mixed Models Analysis
Statistical Analysis 2: Comparison: Prehabilitation; Linear mixed models estimated within-person change in maximum SMIP between baseline and day of surgery; Test type: Superiority; p = 0.734, Mixed Models Analysis — The null hypothesis was rejected a priori if p<.05; Mean Difference (Net) = 10.50, Standard Error of Mean 30.91 — [estimate comment as in outcome 4, analysis 2]
Statistical Analysis 3: Comparison: Prehabilitation; Linear mixed models estimated within-person change in maximum SMIP between baseline and 90 days postop; Test type: Superiority; p = 0.341, Mixed Models Analysis — The null hypothesis was rejected a priori if p<.05; Mean Difference (Net) = 21.07, Standard Error of Mean 22.12 — [estimate comment as in outcome 4, analysis 2]
Statistical Analysis 4: Comparison: Prehabilitation; Linear mixed models estimated within-person change in maximum SMIP between day of surgery and 90 days postop; Test type: Superiority; p = 0.448, Mixed Models Analysis — The null hypothesis was rejected a priori if p<.05; Mean Difference (Net) = 28.55, Standard Error of Mean 37.61 — [estimate comment as in outcome 4, analysis 2]

10. Secondary Outcome: Change in Pulmonary Function Over the Course of Treatment and Recovery: Mean SMIP
Description: Pulmonary function will be measured in terms of mean sustained MIP (SMIP).
Time Frame: Baseline, day of surgery, 90 days postoperatively
Population: All participants that completed the pulmonary function assessments were analyzed at each completed timepoint.
Measure: Mean (Standard Deviation); unit: cm of H2O
Arm/Group | Prehabilitation
Number analyzed (Participants) | 33
cm of H2O
  Baseline Mean SMIP | 364.36 (171.33)
  Day of surgery Mean SMIP: number analyzed (Participants) | 25
  Day of surgery Mean SMIP | 393.86 (185.85)
  90 Day Postop Mean SMIP: number analyzed (Participants) | 22
  90 Day Postop Mean SMIP | 435.94 (202.14)
Statistical Analysis 1: Comparison: Prehabilitation; Linear mixed models estimated overall, within-person change in mean SMIP across all 4 time points; Test type: Superiority; p = 0.419, Mixed Models Analysis
Statistical Analysis 2: Comparison: Prehabilitation; Linear mixed models estimated within-person change in mean SMIP between baseline and day of surgery; Test type: Superiority; p = 0.439, Mixed Models Analysis — The null hypothesis was rejected a priori if p<.05; Mean Difference (Net) = 20.91, Standard Error of Mean 27.03 — [estimate comment as in outcome 4, analysis 2]
Statistical Analysis 3: Comparison: Prehabilitation; Linear mixed models estimated within-person change in mean SMIP between baseline and 90 days postop; Test type: Superiority; p = 0.069, Mixed Models Analysis — The null hypothesis was rejected a priori if p<.05; Mean Difference (Net) = 47.67, Standard Error of Mean 26.19 — [estimate comment as in outcome 4, analysis 2]
Statistical Analysis 4: Comparison: Prehabilitation; Linear mixed models estimated within-person change in mean SMIP between day of surgery and 90 days postop; Test type: Superiority; p = 0.328, Mixed Models Analysis — The null hypothesis was rejected a priori if p<.05; Mean Difference (Net) = 37.11, Standard Error of Mean 37.96 — [estimate comment as in outcome 4, analysis 2]

11. Secondary Outcome: Serum Prealbumin Over the Course of Treatment and Recovery
Description: Higher levels indicate greater levels of protein. Lower levels indicate the potential of inflammation. normal range is 18-41, Below 18 is lower than normal, above 41 is higher than normal
Time Frame: Baseline, day of surgery, 90 days postoperatively
Population: All participants that completed the blood draw were analyzed at each completed timepoint. Additionally, there was an error in the lab when processing the blood samples, this caused many samples to be evaluated incorrectly. Only correctly analyzed labs were included in this analysis.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Prehabilitation
Number analyzed (Participants) | 23
mg/dL
  Baseline Serum Prealbumin | 26.27 (5.57)
  Day of surgery Serum Prealbumin: number analyzed (Participants) | 18
  Day of surgery Serum Prealbumin | 26.50 (4.52)
  90 Day Postop Serum Prealbumin: number analyzed (Participants) | 15
  90 Day Postop Serum Prealbumin | 25.13 (6.48)
Statistical Analysis 1: Comparison: Prehabilitation; Linear mixed models estimated overall, within-person change in serum prealbumin across all 4 time points; Test type: Superiority; p = 0.196, Mixed Models Analysis
Statistical Analysis 2: Comparison: Prehabilitation; Linear mixed models estimated within-person change in serum prealbumin between baseline and day of surgery; Test type: Superiority; p = 0.562, Mixed Models Analysis — The null hypothesis was rejected a priori if p<.05; Mean Difference (Net) = -0.11, Standard Error of Mean 0.19 — [estimate comment as in outcome 4, analysis 2]
Statistical Analysis 3: Comparison: Prehabilitation; Linear mixed models estimated within-person change in serum prealbumin between baseline and 90 days postop; Test type: Superiority; p = 0.087, Mixed Models Analysis — The null hypothesis was rejected a priori if p<.05; Mean Difference (Net) = -0.42, Standard Error of Mean 0.25 — [estimate comment as in outcome 4, analysis 2]
Statistical Analysis 4: Comparison: Prehabilitation; Linear mixed models estimated within-person change in serum prealbumin between day of surgery and 90 days postop; Test type: Superiority; p = 0.226, Mixed Models Analysis — The null hypothesis was rejected a priori if p<.05; Mean Difference (Net) = -0.28, Standard Error of Mean 0.23 — [estimate comment as in outcome 4, analysis 2]

12. Secondary Outcome: Change in Gait Speed Over the Course of Treatment and Recovery
Description: Gait speed will be measured by using a stopwatch to time how long the patient takes to walk 4 meters
Time Frame: Baseline, day of surgery, 90 days postoperatively
Population: All participants that completed the gait speed assessment were analyzed at each completed timepoint.
Measure: Mean (Standard Deviation); unit: m/s
Arm/Group | Prehabilitation
Number analyzed (Participants) | 33
m/s
  Baseline Gait Speed | 1.16 (0.32)
  Day of surgery Gait Speed: number analyzed (Participants) | 24
  Day of surgery Gait Speed | 1.33 (0.28)
  90 Day Postop Gait Speed: number analyzed (Participants) | 22
  90 Day Postop Gait Speed | 1.36 (0.37)
Statistical Analysis 1: Comparison: Prehabilitation; Linear mixed models estimated overall, within-person change in gait speed across all 4 time points; Test type: Superiority; p = 0.001, Mixed Models Analysis
Statistical Analysis 2: Comparison: Prehabilitation; Linear mixed models estimated within-person change in gait speed between baseline and day of surgery; Test type: Superiority; p = 0.001, Mixed Models Analysis — The null hypothesis was rejected a priori if p<.05; Mean Difference (Net) = 0.12, Standard Error of Mean 0.04 — [estimate comment as in outcome 4, analysis 2]
Statistical Analysis 3: Comparison: Prehabilitation; Linear mixed models estimated within-person change in gait speed between baseline and 90 days postop; Test type: Superiority; p = 0.001, Mixed Models Analysis — The null hypothesis was rejected a priori if p<.05; Mean Difference (Net) = 0.16, Standard Error of Mean 0.05 — [estimate comment as in outcome 4, analysis 2]
Statistical Analysis 4: Comparison: Prehabilitation; Linear mixed models estimated within-person change in gait speed between day of surgery and 90 days postop; Test type: Superiority; p = 0.874, Mixed Models Analysis — The null hypothesis was rejected a priori if p<.05; Mean Difference (Net) = 0.01, Standard Error of Mean 0.05 — [estimate comment as in outcome 4, analysis 2]

13. Secondary Outcome: Change in Short Physical Performance Battery (SPPB) Over the Course of Treatment and Recovery
Description: This standardized outcome measure asks patients to complete several activities that are scored independently and then aggregated into an overall score ranging from 0-12. Higher scores indicate better physical performance.
Time Frame: Baseline, day of surgery, 90 days postoperatively
Population: All participants that completed the SPPB assessments were analyzed at each completed timepoint.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Prehabilitation
Number analyzed (Participants) | 33
score on a scale
  Baseline SPPB: number analyzed (Participants) | 32
  Baseline SPPB | 10.44 (1.74)
  Day of surgery SPPB: number analyzed (Participants) | 24
  Day of surgery SPPB | 10.83 (1.17)
  90 Day Postop SPPB: number analyzed (Participants) | 22
  90 Day Postop SPPB | 10.64 (1.94)
Statistical Analysis 1: Comparison: Prehabilitation; Linear mixed models estimated overall, within-person change in SPPB across all 4 time points; Test type: Superiority; p = 0.854, Mixed Models Analysis
Statistical Analysis 2: Comparison: Prehabilitation; Linear mixed models estimated within-person change in SPPB between baseline and day of surgery; Test type: Superiority; p = 0.298, Mixed Models Analysis — The null hypothesis was rejected a priori if p<.05; Mean Difference (Net) = 0.33, Standard Error of Mean 0.32 — [estimate comment as in outcome 4, analysis 2]
Statistical Analysis 3: Comparison: Prehabilitation; Linear mixed models estimated within-person change in SPPB between baseline and 90 days postop; Test type: Superiority; p = 0.684, Mixed Models Analysis — The null hypothesis was rejected a priori if p<.05; Mean Difference (Net) = 0.13, Standard Error of Mean 0.31 — [estimate comment as in outcome 4, analysis 2]
Statistical Analysis 4: Comparison: Prehabilitation; Linear mixed models estimated within-person change in SPPB between day of surgery and 90 days postop; Test type: Superiority; p = 0.485, Mixed Models Analysis — The null hypothesis was rejected a priori if p<.05; Mean Difference (Net) = -0.23, Standard Error of Mean 0.33 — [estimate comment as in outcome 4, analysis 2]

14. Secondary Outcome: Change in Risk Analysis Index of Frailty (RAI) Over the Course of Treatment and Recovery
Description: This recently published frailty index is assessed by a clinician administered questionnaire. The score and reflects frailty-associated mortality risk ranging from 0-81. Higher scores indicate higher risk for post operative complications and other frailty-related outcomes.
Time Frame: Baseline, day of surgery, 90 days postoperatively
Population: All participants that completed the RAI assessment were analyzed at each completed timepoint.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Prehabilitation
Number analyzed (Participants) | 33
score on a scale
  Baseline RAI | 17.85 (8.92)
  Day of surgery RAI: number analyzed (Participants) | 25
  Day of surgery RAI | 20.40 (8.69)
  90 Day Postop RAI: number analyzed (Participants) | 23
  90 Day Postop RAI | 23.30 (9.16)
Statistical Analysis 1: Comparison: Prehabilitation; Linear mixed models estimated overall, within-person change in RAI across all 4 time points; Test type: Superiority; p = 0.067, Mixed Models Analysis
Statistical Analysis 2: Comparison: Prehabilitation; Linear mixed models estimated within-person change in RAI between baseline and day of surgery; Test type: Superiority; p = 0.089, Mixed Models Analysis — The null hypothesis was rejected a priori if p<.05; Mean Difference (Net) = 2.07, Standard Error of Mean 1.22 — [estimate comment as in outcome 4, analysis 2]
Statistical Analysis 3: Comparison: Prehabilitation; Linear mixed models estimated within-person change in RAI between baseline and 90 days postop; Test type: Superiority; p = 0.006, Mixed Models Analysis — The null hypothesis was rejected a priori if p<.05; Mean Difference (Net) = 4.37, Standard Error of Mean 1.60 — [estimate comment as in outcome 4, analysis 2]
Statistical Analysis 4: Comparison: Prehabilitation; Linear mixed models estimated within-person change in RAI between day of surgery and 90 days postop; Test type: Superiority; p = 0.221, Mixed Models Analysis — The null hypothesis was rejected a priori if p<.05; Mean Difference (Net) = 1.98, Standard Error of Mean 1.62 — [estimate comment as in outcome 4, analysis 2]

15. Secondary Outcome: Change in 7-point Subjective Global Assessment (SGA) of Nutrition Over the Course of Treatment and Recovery
Description: This standardized survey instrument is completed by a trained clinician after assessing a nutrition-specific patient history. The minimum score is 1 and the maximum score is 7. High scores indicate better nourishment.
Time Frame: Baseline, day of surgery, 90 days postoperatively
Population: All participants that completed the Subjective Global Assessment were analyzed at each completed timepoint.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Prehabilitation
Number analyzed (Participants) | 26
score on a scale
  Baseline SGA | 6.04 (0.60)
  Day of Surgery SGA: number analyzed (Participants) | 19
  Day of Surgery SGA | 6.00 (0.33)
  90 Day Postop SGA: number analyzed (Participants) | 21
  90 Day Postop SGA | 5.95 (0.59)
Statistical Analysis 1: Comparison: Prehabilitation; Linear mixed models estimated overall, within-person change in SGA across all 4 time points; Test type: Superiority; p = 0.860, Mixed Models Analysis
Statistical Analysis 2: Comparison: Prehabilitation; Linear mixed models estimated within-person change in SGA between baseline and day of surgery; Test type: Superiority; p = 0.410, Mixed Models Analysis — The null hypothesis was rejected a priori if p<.05; Mean Difference (Net) = -0.10, Standard Error of Mean 0.12 — [estimate comment as in outcome 4, analysis 2]
Statistical Analysis 3: Comparison: Prehabilitation; Linear mixed models estimated within-person change in SGA between baseline and 90 days postop; Test type: Superiority; p = 0.622, Mixed Models Analysis — The null hypothesis was rejected a priori if p<.05; Mean Difference (Net) = -0.09, Standard Error of Mean 0.17 — [estimate comment as in outcome 4, analysis 2]
Statistical Analysis 4: Comparison: Prehabilitation; Linear mixed models estimated within-person change in SGA between day of surgery and 90 days postop; Test type: Superiority; p = 0.757, Mixed Models Analysis — The null hypothesis was rejected a priori if p<.05; Mean Difference (Net) = -0.05, Standard Error of Mean 0.15 — [estimate comment as in outcome 4, analysis 2]

16. Secondary Outcome: Change in 6 Minute Walk Test Over the Course of Treatment and Recovery
Description: This standardized approach measures the distance in meters walked during 6 minutes.
Time Frame: Baseline, day of surgery, 90 days postoperatively
Population: All participants that completed the six minute walk test were analyzed at each completed timepoint.
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Prehabilitation
Number analyzed (Participants) | 32
meters
  Baseline 6 Minute Walk Distance | 366.49 (108.68)
  Day of Surgery 6 Minute Walk Distance: number analyzed (Participants) | 22
  Day of Surgery 6 Minute Walk Distance | 400.33 (101.07)
  90 Day Postop 6 Minute Walk Distance: number analyzed (Participants) | 22
  90 Day Postop 6 Minute Walk Distance | 386.96 (94.70)
Statistical Analysis 1: Comparison: Prehabilitation; Linear mixed models estimated overall, within-person change in 6 Minute Walk Test across all 4 time points; Test type: Superiority; p = 0.362, Mixed Models Analysis
Statistical Analysis 2: Comparison: Prehabilitation; Linear mixed models estimated within-person change in 6 Minute Walk Test between baseline and day of surgery; Test type: Superiority; p = .203, Mixed Models Analysis — The null hypothesis was rejected a priori if p<.05; Mean Difference (Net) = 25.52, Standard Error of Mean 20.06 — [estimate comment as in outcome 4, analysis 2]
Statistical Analysis 3: Comparison: Prehabilitation; Linear mixed models estimated within-person change in 6 Minute Walk Test between baseline and 90 days postop; Test type: Superiority; p = 0.357, Mixed Models Analysis — The null hypothesis was rejected a priori if p<0.05; Mean Difference (Net) = 12.70, Standard Error of Mean 13.77 — [estimate comment as in outcome 4, analysis 2]
Statistical Analysis 4: Comparison: Prehabilitation; Linear mixed models estimated within-person change in 6 Minute Walk Test between day of surgery and 90 days postop; Test type: Superiority; p = 0.163, Mixed Models Analysis — The null hypothesis was rejected a priori if p<0.05; Mean Difference (Net) = 21.48, Standard Error of Mean 15.40 — [estimate comment as in outcome 4, analysis 2]

17. Secondary Outcome: Change in Health Related Quality of Life Over the Course of Treatment and Recovery
Description: Assessment of Quality of Life (AQoL-6D) survey. Scores range from 0 to 1. The higher the score, the better the quality of life.
Time Frame: Baseline, day of surgery, 30-days postoperatively, 90-days postoperatively
Population: All participants that completed all of the AQoL6D assessment were analyzed at each completed timepoint.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Prehabilitation
Number analyzed (Participants) | 25
score on a scale
  Baseline AQoL6D Utility Score | 0.72 (0.16)
  Day of surgery AQoL6D Utility Score: number analyzed (Participants) | 22
  Day of surgery AQoL6D Utility Score | 0.75 (0.13)
  90 Day Postop AQoL6D Utility Score: number analyzed (Participants) | 21
  90 Day Postop AQoL6D Utility Score | 0.77 (0.13)
Statistical Analysis 1: Comparison: Prehabilitation; Linear mixed models estimated overall, within-person change across all 4 time points; Test type: Superiority; p = 0.068, Mixed Models Analysis
Statistical Analysis 2: Comparison: Prehabilitation; Linear mixed models estimated within-person change between baseline and day of surgery; Test type: Superiority; p = 0.043, Mixed Models Analysis — The null hypothesis was rejected a priori if p<.05; Mean Difference (Net) = 0.03, Standard Error of Mean 0.02 — [estimate comment as in outcome 4, analysis 2]
Statistical Analysis 3: Comparison: Prehabilitation; Linear mixed models estimated within-person change between baseline and 90 days postop; Test type: Superiority; p = 0.092, Mixed Models Analysis — The null hypothesis was rejected a priori if p<.05; Mean Difference (Net) = 0.04, Standard Error of Mean 0.02 — [estimate comment as in outcome 4, analysis 2]
Statistical Analysis 4: Comparison: Prehabilitation; Linear mixed models estimated within-person change in mean MEP between day of surgery and 90 days postop; Test type: Superiority; p = 0.292, Mixed Models Analysis; The null hypothesis was rejected a priori if p<.05; Mean Difference (Net) = 0.02, Standard Error of Mean 0.02 — [estimate comment as in outcome 4, analysis 2]

18. Other Pre Specified Outcome: Change in Quality of Surgical Care Over the Course of Treatment and Recovery
Description: Agency for Healthcare Research and Quality (AHRQ) Surgical Care Survey (SCS) total communication section. Values are scored on a 3 point scale where 1 is good and 3 bad
Time Frame: Day of Surgery and 30-days postoperatively
Population: All participants that completed the every question of the AHRQ SCS total communication section assessment were analyzed at each completed timepoint.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Prehabilitation
Number analyzed (Participants) | 25
score on a scale
  Day of surgery Total Communication | 1.08 (0.16)
  30 Day Postop Total Communication: number analyzed (Participants) | 24
  30 Day Postop Total Communication | 1.13 (0.43)
Statistical Analysis 1: Comparison: Prehabilitation; Linear mixed models estimated overall, within-person change across both time points; Test type: Superiority; p = 0.625, Mixed Models Analysis

ADVERSE EVENTS:
Time Frame: Adverse events were collected for each participant, from the time of enrollment, usually 3-6 weeks prior to surgery, to first final follow up, 90 days after surgery. Adverse events were collected over a time period of approximately four months.
Arm/Group | Prehabilitation
All-Cause Mortality (participants affected / at risk) | 0/35
Serious Adverse Events (participants affected / at risk) | 7/35
Other Adverse Events (participants affected / at risk) | 0/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Prehabilitation (N=35)
Orthostatic Hypotension (Blood and lymphatic system disorders) | 1 (1) — Patient described slight chest discomfort and tingling to staff, staff noticed that patient was disoriented.
Suspected ischemic stroke (Vascular disorders) | 1 (1)
Unrelated inpatient hospitalization (General disorders) | 1 (2) — Chest pain, shortness of breath, shaking chills after surgery
Detox (General disorders) | 1 (1) — Inpatient prior to surgery for detox.
Unrelated inpatient hospitalization (Respiratory, thoracic and mediastinal disorders) | 1 (2) — Hospitalization for shortness of breath
Post-operative pain unrealted inpatient hospitalization (Injury, poisoning and procedural complications) | 1 (1)
Second unexpect surgery (Surgical and medical procedures) | 1 (1) — Patient needed a second, unexpected surgery. Unrelated to this protocol.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-07-24): https://cdn.clinicaltrials.gov/large-docs/01/NCT03299101/Prot_SAP_000.pdf